CLINICAL TRIAL: NCT06047782
Title: Impact of Atrial Fibrosis Surface Area on the Occurrence of Atrial Fibrillation in Patients With Ischemic Stroke of Undetermined Origin: a Prospective Cardiac MRI Pilot Study.
Acronym: FIBROSIS-MRI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GUENANCIA FRAVC 2022
Record Dates: First submitted 2023-09-05; First posted 2023-09-21 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Implantation of an Implantable Cardiac Monitor
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cardiac MRI (with contrast agent) — Cardiac MRI with contrast agent

SUMMARY:
Atrial fibrillation is a cardiac arrhythmia most often originating in the left atrium, causing anarchic electrical activity and thus a loss of atrial contraction. This increases the risk of stroke through clot formation in the atrium, but also of heart failure. Atrial fibrillation is a major cause of stroke, accounting for more than 25% of all strokes. In addition, a quarter of ischemic strokes remain without an obvious cause at the end of hospitalization, and it is recommended that atrial fibrillation be detected intensively with long-term heart rhythm recording. Implantable loop recorders can detect 30% of atrial fibrillation cases over the 3-year battery life of these devices, after a stroke of undetermined origin. However, these devices require a small operation to implant them under the skin, and they are expensive.

The hypothesis of this study is that MRI imaging of the left atrium would enable better selection of patients to receive an implantable loop recorder. MRI can quantify the proportion of the left atrium with scar tissue, which is likely to favour the onset of atrial fibrillation. If the results confirm this hypothesis, the number of patients requiring an implantable loop recorder could be reduced, and perhaps an anticoagulation strategy based on MRI data could be introduced.

In addition to the usual follow-up by cardiologists and neurologists, participation in this study involves a cardiac MRI (with contrast agent) within 3 months of the stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has provided free, written and informed consent
* Patient of legal age
* Patient with cryptogenic ischemic stroke within 30 days of inclusion, documented by brain imaging (cerebral angioscan or cerebral MRI)
* Patients scheduled for implantable loop recorder implantation within 3 months of ischemic stroke in search of silent AF:

  * cryptogenic ischemic stroke or stroke with probable cardioembolic cause
  * no history of atrial fibrillation
  * no long-term anticoagulant therapy
  * with life expectancy >12 months

Exclusion Criteria:

* Person not affiliated to national health insurance
* Person under legal protection (curatorship, guardianship)
* Person under court order
* Pregnant, parturient or breast-feeding
* Adult unable to give consent
* Patient diagnosed with AF during stroke assessment
* Patient with a contraindication to MRI or gadolinium injection:

  * Severe renal impairment (<30ml/min Cockroft clearance due to gadolinium injection)
  * Claustrophobia / contraindication to MRI (metal implant not MRI compatible)
  * History of hypersensitivity to gadoteric acid or gadolinium-based contrast agents, and to meglumine
  * Uncontrolled asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Episode of atrial fibrillation (AF) lasting more than 30 seconds on the implantable loop recorder | at 3-year follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France